CLINICAL TRIAL: NCT01203488
Title: Randomized Trial of Vitamin A Supplementation for Extremely-Low-Birth-Weight
Brief Title: Vitamin A Supplementation for Extremely-Low-Birth-Weight Infants
Acronym: Vitamin A
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Jon E. Tyson, Lead Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NICHD-NRN-0015; U10HD021373 (NIH); U10HD027904 (NIH); U01HD019897 (NIH); U10HD027871 (NIH); M01RR006022 (NIH); U10HD027851 (NIH); U10HD027856 (NIH); M01RR000750 (NIH); U10HD027880 (NIH); M01RR000070 (NIH); U10HD021397 (NIH); U10HD021415 (NIH); U10HD021364 (NIH); U10HD027853 (NIH); M01RR008084 (NIH); U10HD034216 (NIH); U10HD021385 (NIH); U10HD034167 (NIH); U10HD027881 (NIH); M01RR000997 (NIH)
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature; Bronchopulmonary Dysplasia; Respiration, Artificial; Respiratory Distress Syndrome, Newborn; Sepsis
Keywords: NICHD Neonatal Research Network; Extremely Low Birth Weight (ELBW); Prematurity; Vitamin A; Chronic Lung Disease
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia; Respiratory Aspiration; Respiratory Distress Syndrome, Newborn; Sepsis | interventions — Vitamin A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Vitamin A group.
  Interventions: Drug: Vitamin A
- Control (Sham Comparator): Sham procedure Control group.
  Interventions: Other: Sham Procedure

INTERVENTIONS:
Drug: Vitamin A — 5,000 IU (0.1 ml) was given on Mondays, Wednesdays, and Fridays for four weeks.
  Arms: Experimental
Other: Sham Procedure — Control infants received a sham procedure rather than placebo injections.
  Arms: Control

SUMMARY:
This multi-site, randomized trial was conducted to determine the safety and effectiveness of a higher dose of vitamin A and determine if this would increase the rate of survival without bronchopulmonary dysplasia (BPD) and reduce the risk of sepsis. Infants with birth weights from 401-1000g and who were on mechanical ventilation or supplemental oxygen at 24-96 hours of age were enrolled. Subjects were randomized to either the Vitamin A or a control group. Infants in the Vitamin A group were given a dose of 5000 IU (0.1 ml) intramuscularly on Mondays, Wednesdays, and Fridays for four weeks. Control infants received a sham procedure rather than placebo injections.

DETAILED DESCRIPTION:
Infants with extremely low birth weights (≤1,000 g) have low plasma and tissue concentrations of vitamin A, and vitamin A deficiency may predispose these infants to chronic lung disease. A meta-analysis of clinical trials of vitamin A supplementation for preterm infants revealed a 17% increase in the rate of survival without chronic lung disease, which approached statistical significance.

This multi-site, randomized trial was conducted to determine the safety and effectiveness of a higher dose of vitamin A than that used in previous trials in extremely-low-birth-weight (ELBW) infants. We hypothesized that vitamin A supplementation would increase the rate of survival without bronchopulmonary dysplasia and reduce the risk of sepsis.

Infants with birth weights from 401-1000g and who received mechanical ventilation or supplemental oxygen at 24-96 hours of age were enrolled. Subjects were randomized to either the vitamin A or a control group. Infants in the Vitamin A group were given a dose of 5000 IU (0.1 ml) intramuscularly on Mondays, Wednesdays, and Fridays for four weeks. Control infants received a sham procedure rather than placebo injections.

Serum vitamin A was measured in a central laboratory at base line and at 28 days in the first 300 infants. On study day 28 (two to three days after the last treatment and immediately after a blood sample was collected), the relative dose-response was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Infants wtih birth weights from 401-1,000g
* Receiving mechanical ventilation or supplemental oxygen at 24-96 hours of age

Exclusion Criteria:

* Major congenital anomalies
* Congenital nonbacterial infection
* Infants diagnosed with a terminal illness (as indicated by a pH below 6.80 or by the presence of hypoxia with bradycardia for more than two hours)
* Infants who were to receive vitamin A in a parenteral fat emulsion or in doses exceeding recommendations for multivitamin preparations

Ages: 24 Hours to 96 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 807 (Actual)
Dates: Start 1996-01; Primary Completion 1997-07 (Actual); Study Completion 1999-07 (Actual)

PRIMARY OUTCOMES:
Chronic lung disease or death | 36 weeks' postmenstrual age
  Chronic lung disease was defined as the need for oxygen at 36 weeks' postmenstrual age.

SECONDARY OUTCOMES:
Sepsis | 5 days
  Sepsis was defined on the basis of a positive blood culture and treatment with antibiotics for at least five days (unless the infant died within five days).

CONTACTS AND LOCATIONS:
Overall Officials: Jon E. Tyson, MD MPH, Study Director — University of Texas Southwestern Medical Center; William Oh, MD, Principal Investigator — Brown University, Women and Infants Hospital; Joel Verter, PhD, Principal Investigator — George Washington University Biostatistics Center; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University; Barbara J. Stoll, MD, Principal Investigator — Emory University; James A. Lemons, MD, Principal Investigator — Indiana University; David K. Stevenson, MD, Principal Investigator — Stanford University; Charles R. Bauer, MD, Study Director — University of Miami; Sheldon B. Korones, MD, Principal Investigator — University of Tennessee; Edward F. Donovan, MD, Principal Investigator — Case Western Reserve University
Locations (11):
- United States (11):
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - George Washington University, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Tennessee, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

REFERENCES:
- [Background] Stark AR, Tyson JE, Hibberd PL. Variation among institutional review boards in evaluating the design of a multicenter randomized trial. J Perinatol. 2010 Mar;30(3):163-9. doi: 10.1038/jp.2009.157. Epub 2009 Oct 1. PMID 19798046
- [Result] Kennedy KA, Stoll BJ, Ehrenkranz RA, Oh W, Wright LL, Stevenson DK, Lemons JA, Sowell A, Mele L, Tyson JE, Verter J. Vitamin A to prevent bronchopulmonary dysplasia in very-low-birth-weight infants: has the dose been too low? The NICHD Neonatal Research Network. Early Hum Dev. 1997 Jul 24;49(1):19-31. doi: 10.1016/s0378-3782(97)01869-0. PMID 9179535
- [Result] Tyson JE, Wright LL, Oh W, Kennedy KA, Mele L, Ehrenkranz RA, Stoll BJ, Lemons JA, Stevenson DK, Bauer CR, Korones SB, Fanaroff AA. Vitamin A supplementation for extremely-low-birth-weight infants. National Institute of Child Health and Human Development Neonatal Research Network. N Engl J Med. 1999 Jun 24;340(25):1962-8. doi: 10.1056/NEJM199906243402505. PMID 10379020
- [Result] Ambalavanan N, Tyson JE, Kennedy KA, Hansen NI, Vohr BR, Wright LL, Carlo WA; National Institute of Child Health and Human Development Neonatal Research Network. Vitamin A supplementation for extremely low birth weight infants: outcome at 18 to 22 months. Pediatrics. 2005 Mar;115(3):e249-54. doi: 10.1542/peds.2004-1812. Epub 2005 Feb 15. PMID 15713907
- [Derived] Rysavy MA, Li L, Tyson JE, Jensen EA, Das A, Ambalavanan N, Laughon MM, Greenberg RG, Patel RM, Pedroza C, Bell EF; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Should Vitamin A Injections to Prevent Bronchopulmonary Dysplasia or Death Be Reserved for High-Risk Infants? Reanalysis of the National Institute of Child Health and Human Development Neonatal Research Network Randomized Trial. J Pediatr. 2021 Sep;236:78-85.e5. doi: 10.1016/j.jpeds.2021.05.022. Epub 2021 May 15. PMID 34004189
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org/